CLINICAL TRIAL: NCT00201500
Title: Left Ventricular and Endothelial Function in Preeclampsia, a Case Control Study
Brief Title: Left Ventricular and Endothelial Function in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: PEETLV
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- preeclampsia: women with preeclampsia
- controls: healthy pregnant women

SUMMARY:
The purpose of this study is (1) to examine whether the left ventricular function is impaired in women with preeclampsia relative to healthy pregnant controls, (2) to examine whether the endothelial function is impaired in women with preeclampsia relative to healthy pregnant controls, and (3) to examine whether there is a post partum impairment in left ventricular and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Case: Clinical diagnosis of preeclampsia,
* Control: Systolic BP <140 mmHg and diastolic BP <90 mmHg

Exclusion Criteria:

* Known hypertension or other cardiovascular disease
* Diabetes/gestational diabetes
* Multiple gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with preeclampsia and women with normotensive pregnancies.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Function | 3 months
Endothelial Function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stig A Slørdahl, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- NTNU, Trondheim, Norway

REFERENCES:
- [Result] Tyldum EV, Backe B, Stoylen A, Slordahl SA. Maternal left ventricular and endothelial functions in preeclampsia. Acta Obstet Gynecol Scand. 2012 May;91(5):566-73. doi: 10.1111/j.1600-0412.2011.01282.x. PMID 21943052